CLINICAL TRIAL: NCT05755451
Title: Natural History of SMA: Long Term Longitudinal Study and Development of a Registry
Brief Title: Natural History of SMA
Acronym: iSMAR
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University of Milan (Other); Istituto Giannina Gaslini (Other); Ospedale Pediatrico Bambin Gesù (Other); University of Messina (Other)
Responsible Party: Sponsor
Other Study IDs: 1894
Record Dates: First submitted 2023-02-08; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Muscular Atrophy, Spinal
Keywords: natural history; spinal muscular atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an investigator initiated observational study with the aim to record several aspects of function, care and adverse events in a large cohort of SMA patients followed longitudinally by using a structured academic disease registry.

DETAILED DESCRIPTION:
This is an observational multicenter retrospective and prospective study involving high quality data collected in 5 academic centers in Italy, the registry aims to

* better understand the natural history of the disease in untreated patients identifying factors that can influence disease progression by combining retrospective and prospective data.
* Describe the patterns of disease progression (in terms of functional measure, adverse events, levels of care, and hospitalization) in treated and untreated patients
* Identify all the patients treated with the available therapies in Italy, providing first line details on epidemiological data in a wider network including all centers recognized as centers for spinal muscular atrophy (SMA) in each region.

As part of the activity clinical evaluators, data manager and sub-investigators are also trained and use common manuals of operation to ensure reliability across the participating centers. The registry provides accurate and reliable information on natural history including results from currently used functional measures. The registry also includes information on supportive care, hospitalization and adverse events.

Details of the electronic clinical file record including data assembly and the platform used are available as part of a peer reviewed paper

ELIGIBILITY:
Inclusion Criteria:

all patients

Exclusion Criteria:

if enrolled in clinical trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all pèatients with mutations in the SMN1 gene
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2033-12-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
motor function | 15 years
  functional scales Hammersmith Functional motor scale, (minimum score 0, maximum score 74 indicating best performance

SECONDARY OUTCOMES:
respiratory function | 15 years
  Forced Vital Capacity, need for ventilatory support
nutrition | 15 years
  need for nutritional support using Oral and Swallowing Abilities Tool (OrSAT) with a minimum score of 0 and a maximum score of 12 indicating best performance

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Mercuri, MD, Principal Investigator — F Policlinico Gemelli IRCCS
Locations (5):
- Italy (5):
  - Istituto Gaslini, Genova
  - Nemo Sud, Messina
  - Centro Clinico nemo, Milan
  - Ospedale Bambino gesu, Rome
  - Policlinico gemelli, Rome

IPD SHARING:
Plan to Share IPD: No
aggregate data only